CLINICAL TRIAL: NCT02576093
Title: First-in-human, Single Center, Combined SAD/MAD, Double-blind, Placebo-controlled, Half-side Comparison Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of 0.1%, 0.3% and 1% WOL071-007-containing Formulations in Atopic Dermatitis Patients
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of WOL071-007 in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KOR1-14/2013
Record Dates: First submitted 2015-09-04; First posted 2015-10-15 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.1% WOL071-007 (Experimental): Formulation containing 0.1% WOL071-007 for topical application
  Interventions: Drug: 0.1% WOL071-007
- 0.3% WOL071-007 (Experimental): Formulation containing 0.3% WOL071-007 for topical application
  Interventions: Drug: 0.3% WOL071-007
- 1.0% WOL071-007 (Experimental): Formulation containing 1.0% WOL071-007 for topical application
  Interventions: Drug: 1.0% WOL071-007
- WOL071-007 Placebo (Placebo Comparator): Formulation containing Placebo of WOL071-007 for topical application
  Interventions: Drug: Placebo of WOL071-007

INTERVENTIONS:
Drug: 0.1% WOL071-007 — Application of approximately 2 mg cream/cm² skin to a defined surface area. SAD part: Single application to ≤ 100 cm² of non-lesional or lesional skin; MAD part: Multiple application (6 Days) to 2000 cm² of lesional and non-lesional skin.
  Arms: 0.1% WOL071-007
Drug: 0.3% WOL071-007 — Application of approximately 2 mg cream/cm² skin to a defined surface area. SAD part: Single application to ≤ 100 cm² of non-lesional or lesional skin; MAD part: Multiple application (6 Days) to 2000 cm² of lesional and non-lesional skin.
  Arms: 0.3% WOL071-007
Drug: 1.0% WOL071-007 — Application of approximately 2 mg cream/cm² skin to a defined surface area. SAD part: Single application to ≤ 100 cm² of non-lesional or lesional skin; MAD part: Multiple application (6 Days) to 2000 cm² of lesional and non-lesional skin.
  Arms: 1.0% WOL071-007
Drug: Placebo of WOL071-007 — Application of approximately 2 mg cream/cm² skin to a defined surface area. SAD part: Single application to ≤ 100 cm² of non-lesional or lesional skin; MAD part: Multiple application (6 Days) to 2000 cm² of lesional and non-lesional skin.
  Arms: WOL071-007 Placebo

SUMMARY:
Purpose of the study is the local tolerability and systemic safety of a novel k-opioid receptor agonist proven to inhibit inflammation and pruritus in preclinical model of dermatitis.

Three concentrations of WOL071-007 and placebo will be applied to patients with AD in a first-in-human, single-center, combined single/multiple ascending dose (SAD/MAD), double-blind, placebo-controlled, half-side comparison (MAD part only) study. The IMP will be applied occlusively to lesional or non-lesional skin. In the SAD part 24 subjects will receive the IMP for 2 days. In the MAD part, 30 hospitalized subjects will receive the IMP for 6 days. Study objectives are the safety and tolerability as well as (MAD part only) the pharmacokinetics and efficacy of WOL071-007.

DETAILED DESCRIPTION:
Three concentrations of the Investigational Medicinal Product (IMP) WOL071-007 (= active IMP) or placebo will be applied to patients with a clinical diagnosis of atopic dermatitis at screening with an Investigator's Global Dermatitis Assessment (IGADA) score of 1 or 2 (mild to moderate) and/or a local SCORing Atopic Dermatitis (SCORAD) ≤12.

Each dose level cohort will begin with 2 sentinel patients: 1 patient randomized to receive active IMP and the other patient randomized to receive placebo only. From the remaining patients 1 patient will be randomized to receive placebo.

In the Single Ascending Dose (SAD) part of the study the active IMP or placebo will be applied to a defined surface area of ≤ 100 cm² of non-lesional skin (Day 1) or lesional skin (Day 2) for about 22 hours and the patients will remain in the study center for at least 6 hours after dosing.

In the Multiple Ascending Dose (MAD) part placebo or test product + placebo (half-side comparison) will be administered up to 24 hours to achieve a defined surface area of approximately 2000 cm² in total (10% Body Surface Area) for each dose level cohort. A Data Safety Monitoring Board will review the data and recommend continuation following each dose level cohort.

Primary criteria for evaluation are safety assessments, e.g. by Adverse Event (AE) recording, and assessments of the local tolerability (by scoring of local symptoms) as well as of the systemic tolerability (e.g. by blood tests and neurological examination) of WOL071-007. In the MAD part additionally pharmacokinetics will be measured and as secondary parameter local efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, including acceptance of biopsies.
* Male / female.
* Age between 18 and 75 years.
* Body weight between 60 and 130 kg for males and between50 and 110 kg for females. In addition the Body Mass Index (BMI) range limit of 19 - 32 kg/m² (both inclusive) is applicable.
* Lesional skin (at least 50 cm²) anywhere on the body (non-hairy skin) (SAD part only).
* Score of ≥40mm on all screening pruritus visual analogue scale (vas) assessments (average and worst over the last 24 hours and current itch) (MAD part only).
* Stable disease for ≥7 days prior to screening (MAD part only).
* Eczema on the right and left crook of the arms, or in the hollow of the knees (MAD part only).

Exclusion Criteria:

* Absence of written informed consent upon enrolment.
* Atopic dermatitis only affecting the head or scalp. Unstable or actively infected atopic dermatitis.
* Patients with severe atopic dermatitis (IGADA score >2 or local SCORAD >12).
* Concomitant dermatologic or medical condition(s) assessed by the investigator which may interfere with the investigator's ability to evaluate the patient's response to the study drug.
* Patients who have received monoclonal antibody therapy for their atopic dermatitis in the 4 months prior to the start of study treatment.
* Patients who have used systemic immunosuppressive drugs, corticosteroids or received puva therapy in the 4 weeks prior to starting study treatment, or are scheduled to start these treatments during the study period.
* Patients who have used topical immunomodulators (such as pimecrolimus, tacrolimus) within 1 week of starting study treatment or are scheduled to start these treatments during the study period.
* Patients who have used topical corticosteroids from who group II, III or IV, or other treatments for atopic dermatitis, including wet wraps, within 1 week prior to starting study treatment or are likely to require treatment with these medications during the study period of the SAD and MAD parts and from day 7 until day 14 of the MAD part.
* Patients who are unable to abstain from using emollients in the target imp (verum and placebo) assessment areas from day -3 until day 4 during the SAD part and from day -3 until day 14 during the MAD part.
* Patients who are using any concomitant medication(s), e.g. antihistamines, psychotropic drugs, immunosuppressive drugs, and immunologic drugs that, in the investigators' opinion, could affect the patient's atopic dermatitis or pruritus. Patients using such medications may be included, at the investigators discretion, if they have been stable on treatment for at least 1 month prior to the start of study treatment and no changes to these medications are planned during the study period.
* Patients undergoing ultraviolet A or B (UVA or UVB) therapy in the 2 weeks prior to starting study treatment or during the study period.
* Planned exposure of affected areas to excessive sunlight.
* Patients with any of the liver function tests (aspartate aminotransferase [ast], alanine aminotransferase [alt], alkaline phosphatase [alp], gamma-glutamyl-transferase [ggt]) >2.0 x upper limit of normal, or with any clinically significant abnormal safety laboratory tests.
* Patients who are receiving any investigational drug or who have taken part in a clinical study with an investigational drug within three months prior to the start of study treatment.
* History of hypersensitivity and/or idiosyncrasy to any of the test compounds or excipients employed in this study.
* Patients who are HIV-seropositive.
* History or presence of alcohol or substance abuse.
* Regular smokers (more than 20 cigarettes or 5 cigars per day).
* Clinically relevant physical abnormalities, medical conditions or clinical laboratory test results e.g. gastrointestinal, renal, hepatic, pulmonary, cardiac, hematological, endocrinological, neurological, or psychiatric conditions.
* Clinically relevant symptoms (other than those in the inclusion criteria) within two weeks prior to the start of the study.
* History of blood loss exceeding 450 ml (including blood donations) within 1 month before the study.
* History of clinically relevant jaundice (exceptions: completely healed hepatitis a, new-born infant's jaundice).
* Clinically relevant abnormalities in the 12-lead electrocardiogram (ECG) with marked baseline prolongation (QT/QTC, QTC interval > 500 msec) [QTC=corrected QT interval].
* Relevant systemic disease history, either past with sequel, or present, on physical examination.
* any condition (surgical or medical) which may affect absorption, distribution, metabolism and/or excretion of the drug.
* Known history of either an acute or chronic allergy requiring medical therapy.
* Intake of any medical treatment, e.g. antihistamines, including over the counter products, within one week before start of treatment or during the study (with the exception of dietary supplements such as iodine or fluoride in physiological doses), which could interfere with study medication in the opinion of the investigator.
* Not willing to give consent for transmission of personal "pseudonymity" data.
* Not willing and able to use a contraceptive method. Reliable methods for women are double barrier methods including hormonal contraceptives, surgical intervention (e.g. tubal ligation), intrauterine device (IUD) or sexual abstinence, e.g. condoms used plus spermicide or oral contraceptives. Women must use reliable methods from 6 weeks before the first administration of test product until 3 weeks after the last administration of the study medication. Men must use reliable methods from 3 weeks before the first administration of test product until 3 months after the last administration of the study medication. Reliable methods for men are condoms and sexual abstinence.
* For females: pregnancy or lactation.
* Patients who are unable to comply with the requirements of the study or who in the opinion of the investigator should not participate in the study.
* Regular consumption of large amounts of caffeine-containing beverages which, in the opinion of the investigator, could interfere with study procedures.
* Subject is a vulnerable subject (e.g. kept in detention).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety of WOL071-007 by recording adverse events (AEs) and other safety parameters over the Study Period | SAD part: 2 days; MAD part: 7 days
  Number of participants with AEs related to treatment and/or abnormal vital signs (blood pressure, pulse and temperature), monitored on each study day.
Local tolerability over the Study Period | SAD part: 2 days; MAD part: 7 days
  Number of participants with a change in at least one item of local tolerability scores (erythema, edema, vesiculation, oozing, scaling, cracking or crazing, scabbing, papules, reaction spreading outside area of application, glazing, burning or stinging), monitored on each study day.
Systemic Tolerability over the Study Period | SAD part: 2 days; MAD part: 7 days
  Number of participants with results from neurological examination other than normal (covering possible central and peripheral neurological disorders) and/or with abnormal safety laboratory values (standard hematology, blood chemistry), monitored on each study day.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) over the Treatment Period (MAD part only) | 6 days
  Determined from 24h blood sampling (pre-dose and after 1h, 2h, 4h, 6h, 8h and 24h) on days 1, 3, 4, 5 and 6; Plasma concentration-time data will be summarized by treatment with descriptive statistics and mean and individual plasma concentration-time curves will be plotted.
Change in Local Pruritus Intensity over the Study Period (MAD part only) | 7 days
  To be assessed by the patient (self-reporting) using the visual analogue scale, monitored on each study day.
Change in Atopic Dermatitis Severity assessed by Eczema Area and Severity Index (EASI) over the Study Period (MAD part only) | 7 days
  To be assessed at the treated skin area and by the change from baseline.
Change in Atopic Dermatitis Severity assessed by IGADA scores over the Study Period (MAD part only) | 7 days
  To be assessed at the treated skin area and by the change from baseline.
Change in Atopic Dermatitis Severity assessed by local SCORAD over the Study Period (MAD part only) | 7 days
  To be assessed at the treated skin area and by the change from baseline, monitored on each study day.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Abels, MD, Study Director — Dr. August Wolff GmbH & Co. KG Arzneimittel; Georg Golor, MD, Principal Investigator — Parexel GmbH
Locations (1):
- PAREXEL International GmbH Early Phase, Berlin, State of Berlin, Germany